CLINICAL TRIAL: NCT01609296
Title: The IN.PACT Global Clinical Study for the Treatment of Comprehensive Superficial Femoral and/or Popliteal Artery Lesions Using the IN.PACT Admiral™ Drug-Eluting Balloon.
Brief Title: IN.PACT Global Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10048613
Record Dates: First submitted 2012-05-24; First posted 2012-05-31 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Drug coated balloon; Superficial Femoral Artery; Popliteal Femoral Artery; Atherosclerosis; Drug eluting balloon
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IN.PACT Admiral DEB (Experimental): The subjects in this trial will be treated with the IN.PACT Admiral™ percutaneous transluminal angioplasty (PTA) paclitaxel drug eluting balloon (hereinafter referred as "IN.PACT Admiral™ DEB")manufactured by Medtronic. The IN.PACT Admiral™ is a CE (Conformité Europeénne, European Confirmity) marked medical device utilized within its intended use in the IN.PACT Global trial.
  Interventions: Device: IN.PACT Admiral™ Drug Eluting Balloon

INTERVENTIONS:
Device: IN.PACT Admiral™ Drug Eluting Balloon — IN.PACT Admiral™ percutaneous transluminal angioplasty (PTA) paclitaxel drug eluting balloon.

SUMMARY:
The purpose of this study is to collect safety and efficacy data on the IN.PACT Admiral™ Drug Eluting Balloon (DEB) in treatment of atherosclerotic disease in the superficial femoral and/or popliteal arteries in a "real world" patient population.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) commonly results from progressive narrowing of the arteries in the lower extremities, usually due to atherosclerosis. Progression of PAD can result in critical limb ischemia (CLI), manifested by ischemic pain at rest or in the breakdown of the skin, resulting in ulcers or gangrene which ultimately may lead to amputation and death.

The IN.PACT Global Clinical Study aims to expand and understand the safety and efficacy data on the IN.PACT Admiral™ DEB in a real world population of subjects with intermittent claudication and/or rest pain (Rutherford class 2-3-4) due to obstructive disease of the superficial femoral and/or popliteal arteries.

ELIGIBILITY:
General inclusion Criteria:

* Age ≥ 18 years or minimum age as required by local regulations.
* Subject with documented diagnosis of peripheral arterial disease (PAD) in the superficial femoral artery (SFA) and/or popliteal artery (PA) (including P1, P2, P3) classified as Rutherford class 2-3-4.
* Angiographically documented single or multiple lesions/occlusions (de novo or re-stenotic lesion(s) or in-stent restenosis) within the target vessels with a minimum lesion length of 2 cm including bilateral disease if both limbs are treated within 35 days.

General exclusion Criteria:

* High probability of non-adherence to Clinical Investigation Protocol follow-up requirements.
* Failure to successfully cross the target lesion with a guide wire (successful crossing means tip of the guide wire distal to the target lesion in the absence of flow limiting dissections or perforations).
* Lesion within or adjacent to an aneurysm or presence of a popliteal aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1535 (Actual)
Dates: Start 2012-05; Primary Completion 2016-04 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — Klinikum Rosenheim; Gary Ansel, MD, Principal Investigator — MidOhio Cardiology and Vascular Consultants; Marc Bosiers, MD, Principal Investigator — AZ Sint Blasius; Do-Dai Do, MD, Principal Investigator — Swiss Cardiovascular Center, Inselspital; Peter Gaines, MD, Principal Investigator — Sheffield Vascular Institute; Alvaro Razuk, MD, Principal Investigator — Faculdade de Ciências Médicas da Santa Casa de Sao Paulo
Locations (65):
- Argentina (2):
  - Fundación Favaloro, Buenos Aires
  - Clinica La Sagrada Familia, Bueos Aires
- Royal Prince Alfred Hospital, Sydney, Australia
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Landesklinikum Thermenregion Mödling, Mödling
- Belgium (7):
  - Onze-Lieve-Vrouwziekenuis, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - AZ St. Blasius, Dendermonde
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost Limburg - Campus St.-Jan, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Regionaal Ziekenhuis Heilig Hart, Tienen
- Canada (2):
  - Centre hospitalier universitaire Sherbrooke (CHUS), Sherbrooke
  - Toronto General Hospital, Toronto
- Colombia (2):
  - Clinica Santa Maria, Medellín
  - Clinica Medilaser Neiva, Neiva
- Faculty Hospital Hradec Kralove, Hradec Králové, Czechia
- Egypt (2):
  - As-Salam International Hospital, Cairo
  - Egypt Air Hospital, Cairo
- Helsingin Seudun Yliopistollinen Keskussairaala, Helsinki, Finland
- France (2):
  - Group Hospitalier Pellegrin - CHU, Bordeaux
  - Les Hospitaux Universitaires de Strasbourg, Strasbourg
- Germany (9):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Augusta Krankenhaus, Düsseldorf
  - Augusta-Krankenhaus, Düsseldorf
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Leipzig AoR, Leipzig
  - Park-Krankenhaus Leipzig, Leipzig
  - St. Franziskus Hospital GmbH, Münster
  - RoMed Klinikum Rosenheim, Rosenheim
  - Universitätsklinikum Tübingen, Tübingen
- University Hospital of Patras, Pátrai, Greece
- Hungary (2):
  - Semmelweis University, Budapest
  - Bacs Kiskun Megyei Korhaz, Kecskemét
- Israel (2):
  - Carmel Medical Centre, Haifa
  - Rabin Medical Center - Beilison Hospital, Petah Tikva
- Italy (3):
  - Policlinico Vittorio Emanuele, Catania
  - Maria Eleonora Hospital, Palermo
  - Policlinico Gemelli, Rome
- Kaunas Mecial University Clinic, Kaunas, Lithuania
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Ziekenhuis, Arnhem
  - Catharina Ziekenhuis, Eindhoven
  - Sint Antonius Hospital, Nieuwegein
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (2):
  - Euromedic Medical Center, Katowice
  - Samodzielny Publiczny Szpital Kliniczny Nr 2, Szczecin
- Hospital Santa Marta, Lisbon, Portugal
- City Clinical Hospital named after M.E. Zhadkevich, Moscow, Russia
- Changi General Hospital, Singapore, Singapore
- Slovakia (3):
  - Stredoslovensky ustav srdcovych a cievnych chorob (SUSCCH), Banská Bystrica
  - Národný ústav srdcových a cievnych chorôb a.s. (NUSCH), Bratislava
  - Východoslovenský ústav srdcových a cievnych chorôb, a.s.(VUSH), Košice
- University Medical Centre Maribor, Maribor, Slovenia
- South Korea (5):
  - Severence Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
- Karolinska Universitetssjukhuset, Solna, Sweden
- Switzerland (3):
  - Inselspital - Universitätsspial Bern, Bern
  - Hopital Cantonal HFR, Fribourg
  - Kantonspital Luzern, Lucerne
- United Kingdom (2):
  - Manchester Royal Infirmary, Manchester
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ansel GM, Brodmann M, Rocha-Singh KJ, Menk JS, Zeller T; IN.PACT Global Study Investigators. Five-Year Safety and Effectiveness of Paclitaxel Drug-Coated Balloons Alone or With Provisional Bare Metal Stenting for Real-World Femoropopliteal Lesions: IN.PACT Global Study Subgroup Analysis. Circ Cardiovasc Interv. 2024 Feb;17(2):e013084. doi: 10.1161/CIRCINTERVENTIONS.123.013084. Epub 2024 Feb 13. PMID 38348677
- [Derived] Krishnan P, Farhan S, Schneider P, Kamran H, Iida O, Brodmann M, Micari A, Sachar R, Urasawa K, Scheinert D, Ando K, Tarricone A, Doros G, Tepe G, Yokoi H, Laird J, Zeller T. Determinants of Drug-Coated Balloon Failure in Patients Undergoing Femoropopliteal Arterial Intervention. J Am Coll Cardiol. 2022 Sep 27;80(13):1241-1250. doi: 10.1016/j.jacc.2022.06.043. PMID 36137674
- [Derived] Brodmann M, Lansink W, Guetl K, Micari A, Menk J, Zeller T. Long-Term Outcomes of the 150 mm Drug-Coated Balloon Cohort from the IN.PACT Global Study. Cardiovasc Intervent Radiol. 2022 Sep;45(9):1276-1287. doi: 10.1007/s00270-022-03214-y. Epub 2022 Jul 21. PMID 35864209
- [Derived] Zeller T, Brodmann M, Ansel GM, Scheinert D, Choi D, Tepe G, Menk J, Micari A. Paclitaxel-coated balloons for femoropopliteal peripheral arterial disease: final five-year results of the IN.PACT Global Study. EuroIntervention. 2022 Dec 2;18(11):e940-e948. doi: 10.4244/EIJ-D-21-01098. PMID 35635160
- [Derived] Torsello G, Stavroulakis K, Brodmann M, Micari A, Tepe G, Veroux P, Benko A, Choi D, Vermassen FEG, Jaff MR, Guo J, Dobranszki R, Zeller T; IN.PACT Global Investigators. Three-Year Sustained Clinical Efficacy of Drug-Coated Balloon Angioplasty in a Real-World Femoropopliteal Cohort. J Endovasc Ther. 2020 Oct;27(5):693-705. doi: 10.1177/1526602820931477. Epub 2020 Jun 25. PMID 32583749
- [Derived] Shishehbor MH, Schneider PA, Zeller T, Razavi MK, Laird JR, Wang H, Tieche C, Parikh SA, Iida O, Jaff MR. Total IN.PACT drug-coated balloon initiative reporting pooled imaging and propensity-matched cohorts. J Vasc Surg. 2019 Oct;70(4):1177-1191.e9. doi: 10.1016/j.jvs.2019.02.030. PMID 31543165
- [Derived] Reijnen MMPJ, van Wijck I, Zeller T, Micari A, Veroux P, Keirse K, Lee SW, Li P, Voulgaraki D, Holewijn S. Outcomes After Drug-Coated Balloon Treatment of Femoropopliteal Lesions in Patients With Critical Limb Ischemia: A Post Hoc Analysis From the IN.PACT Global Study. J Endovasc Ther. 2019 Jun;26(3):305-315. doi: 10.1177/1526602819839044. Epub 2019 Apr 1. PMID 30931726
- [Derived] Tepe G, Micari A, Keirse K, Zeller T, Scheinert D, Li P, Schmahl R, Jaff MR; IN.PACT Global Study Investigators. Drug-Coated Balloon Treatment for Femoropopliteal Artery Disease: The Chronic Total Occlusion Cohort in the IN.PACT Global Study. JACC Cardiovasc Interv. 2019 Mar 11;12(5):484-493. doi: 10.1016/j.jcin.2018.12.004. PMID 30846089
- [Derived] Schneider PA, Laird JR, Doros G, Gao Q, Ansel G, Brodmann M, Micari A, Shishehbor MH, Tepe G, Zeller T. Mortality Not Correlated With Paclitaxel Exposure: An Independent Patient-Level Meta-Analysis of a Drug-Coated Balloon. J Am Coll Cardiol. 2019 May 28;73(20):2550-2563. doi: 10.1016/j.jacc.2019.01.013. Epub 2019 Jan 25. PMID 30690141
- [Derived] Zeller T, Brodmann M, Micari A, Keirse K, Peeters P, Tepe G, Scheinert D, Jaff MR, Rocha-Singh KJ, Li P, Schmahl R, Ansel GM; IN.PACT Global Study Investigators. Drug-Coated Balloon Treatment of Femoropopliteal Lesions for Patients With Intermittent Claudication and Ischemic Rest Pain. Circ Cardiovasc Interv. 2019 Jan;12(1):e007730. doi: 10.1161/CIRCINTERVENTIONS.118.007730. No abstract available. PMID 30630355
- [Derived] Banerjee S, Khalili H. Drug-Coated Balloon for Long Femoropopliteal Lesions. Circ Cardiovasc Interv. 2018 Oct;11(10):e007084. doi: 10.1161/CIRCINTERVENTIONS.118.007084. No abstract available. PMID 30354645
- [Derived] Scheinert D, Micari A, Brodmann M, Tepe G, Peeters P, Jaff MR, Wang H, Schmahl R, Zeller T; IN.PACT Global Study Investigators. Drug-Coated Balloon Treatment for Femoropopliteal Artery Disease. Circ Cardiovasc Interv. 2018 Oct;11(10):e005654. doi: 10.1161/CIRCINTERVENTIONS.117.005654. PMID 30354636
- [Derived] Ansel GM, Brodmann M, Keirse K, Micari A, Jaff MR, Rocha-Singh K, Fernandez EJ, Wang H, Zeller T; IN.PACT Global Study Investigators. Drug-Coated Balloon Treatment of Femoropopliteal Lesions Typically Excluded From Clinical Trials: 12-Month Findings From the IN.PACT Global Study. J Endovasc Ther. 2018 Dec;25(6):673-682. doi: 10.1177/1526602818803119. Epub 2018 Oct 3. PMID 30280648
- [Derived] Micari A, Brodmann M, Keirse K, Peeters P, Tepe G, Frost M, Wang H, Zeller T; IN.PACT Global Study Investigators. Drug-Coated Balloon Treatment of Femoropopliteal Lesions for Patients With Intermittent Claudication and Ischemic Rest Pain: 2-Year Results From the IN.PACT Global Study. JACC Cardiovasc Interv. 2018 May 28;11(10):945-953. doi: 10.1016/j.jcin.2018.02.019. PMID 29798770

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinical Cohort ITT
Started | 1406
Completed | 918
Not Completed | 488
Not completed — Death | 253
Not completed — Withdrawal by Subject | 151
Not completed — Lost to Follow-up | 21
Not completed — Exit reason other than withdrawal, death or lost to follow up | 35
Not completed — missed visit but known to be alive | 28

BASELINE CHARACTERISTICS:
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1406
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to missing data number analyzed for age differs from overall number of participants
  years
    number analyzed (Participants) | 1396
    (all) | 68.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 453
  Male | 953

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cohort ITT - Primary Effectiveness Endpoint
Description: Freedom from clinically-driven target lesion revascularization (TLR) within 12 months post-index procedure, which is defined as: • Any re-intervention within the target lesion(s) due to symptoms or drop of ABI ≥ 20% or > 0.15 when compared to post-index procedure baseline ABI.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1361
Participants | 1263

2. Primary Outcome: Clinical Cohort ITT - Primary Safety Endpoint
Description: A composite of freedom from device- and procedure-related mortality through 30 days, freedom from major target limb amputation and TLR within 12 months post-index procedure.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1361
Participants | 1254

3. Primary Outcome: Imaging Cohort ITT - Primary Effectiveness Endpoint
Description: Primary Patency within 12 months post-index procedure, which is defined as:
  * Freedom from clinically-driven TLR and
  * Freedom from restenosis as determined by DUS Peak Systolic Velocity Ratio (PSVR) ≤ 2.4.
    * Restenosis determined by either PSVR >2.4 as assessed by an independent DUS core lab or >50% stenosis as assessed by an independent angiographic core lab.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Imaging Cohort ITT
Number analyzed (Participants) | 323
Participants | 217

4. Primary Outcome: 150mm DEB ITT Cohort - Primary Effectiveness Endpoint
Description: as for outcome 1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 106

5. Secondary Outcome: Clinical Cohort ITT - MAEs
Description: MAE (Major Adverse Events) is defined as all-cause mortality, clinically-driven TVR (Target Vessel Revascularization), major target limb amputation, thrombosis at the target lesion site.
Time Frame: 12 months
Population: Event rates are based on number of evaluable subjects - subjects with at least one MAE event within 360-day or subjects without any MAE event but had at least 300 days of clinical follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1361
Participants
  All MAE | 161
  All cause death | 49
  CD-TVR | 107
  Major Target Limb Amputation | 3
  Thrombosis at Target Lesion Site | 38

6. Secondary Outcome: Clinical Cohort ITT - TLR
Description: Any Target lesion revascularisation
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1361
Participants | 101

7. Secondary Outcome: Clinical Cohort ITT - TVR
Description: Any Target vessel revascularisation
Time Frame: 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1361
Participants | 110

8. Secondary Outcome: Clinical Cohort ITT - Device Success
Description: Device success is defined as successful delivery, balloon inflation and deflation and retrieval of the intact study device without burst below the rated burst pressure (RBP)
Time Frame: Index-procedure
Measure: Count of Units; unit: Admiral™ Drug-Eluting Balloon
Units Other Than Participants: Admiral™ Drug-Eluting Balloon
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1406
Number analyzed (Admiral™ Drug-Eluting Balloon) | 3006
Admiral™ Drug-Eluting Balloon | 2988

9. Secondary Outcome: Clinical Cohort ITT - Clinical Success
Description: Clinical success is defined as procedural success without procedural complications (mortality, major target limb amputation, thrombosis of the target lesion, or TVR) prior to discharge
Time Frame: prior to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1396
Participants | 1376

10. Secondary Outcome: Clinical Cohort ITT - MAEs
Description: MAE (Major Adverse Events) is defined as all-cause mortality, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site.
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Cohort ITT: Death, Major Target Limb Amputation, Clinically-driven TVR, Thrombosis
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1215
Participants
  MAEs | 589
  Deaths | 244
  CD-TVR | 381
  Major Target Limb Amputation | 19
  Thrombosis At Target Lesion Site | 73

11. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TLR
Description: Clinically-driven TLR is defined as any re-intervention at the target lesion due to symptoms or drop of ABI of ≥ 20% or > 0.15 when compared to post-index procedure baseline ABI.
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1215
Participants | 366

12. Secondary Outcome: Clinical Cohort ITT - TVR
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1215
Participants | 390

13. Secondary Outcome: Clinical Cohort ITT - TLR
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1215
Participants | 374

14. Secondary Outcome: Clinical Cohort ITT - Time to First Clinically-driven TLR (Days)
Time Frame: 60 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 366
Days | 669.2 (462.5)

15. Secondary Outcome: Clinical Cohort ITT - MAEs
Description: Major Adverse Events (MAE) defined as all-cause death, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site at 30 days.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1403
Participants
  MAEs | 19
  Death | 3
  CD-TVR | 13
  Major Target Limb Amputation | 0
  Thrombosis at Target Lesion Site | 14

16. Secondary Outcome: Clinical Cohort ITT - MAEs
Description: MAE is defined as all-cause mortality, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1386
Participants
  MAEs | 82
  Death | 23
  CD-TVR | 54
  Major Target Limb Amputation | 3
  Thrombosis at Target Lesion Site | 28

17. Secondary Outcome: Clinical Cohort ITT - MAEs
Description: as for outcome 16
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1313
Participants
  MAEs | 325
  Deaths | 101
  CD-TVR | 224
  Major Target Limb Amputation | 9
  Thrombosis at Target Lesion Site | 57

18. Secondary Outcome: Clinical Cohort ITT - MAEs
Description: as for outcome 16
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1277
Participants
  MAEs | 438
  All cause deaths | 147
  CD-TVR | 298
  Major Target Limb Amputation | 12
  Thrombosis at Target Lesion Site | 71

19. Secondary Outcome: Clinical Cohort ITT - MAEs
Description: as for outcome 16
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1242
Participants
  MAEs | 517
  All cause deaths | 196
  CD-TVR | 342
  Major Target Limb Amputation | 15
  Thrombosis at Target Lesion Site | 71

20. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1403
Participants | 13

21. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1386
Participants | 51

22. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1313
Participants | 214

23. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1277
Participants | 288

24. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1242
Participants | 331

25. Secondary Outcome: Clinical Cohort ITT - TLR
Description: Any Target lesion revascularisation
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1386
Participants | 53

26. Secondary Outcome: Clinical Cohort ITT - TLR
Description: Any Target lesion revascularisation
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1313
Participants | 218

27. Secondary Outcome: Clinical Cohort ITT - TLR
Description: Any Target lesion revascularisation
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1277
Participants | 294

28. Secondary Outcome: Clinical Cohort ITT - TLR
Description: Any Target lesion revascularisation
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1242
Participants | 338

29. Secondary Outcome: Clinical Cohort ITT - TVR
Description: Any Target lesion revascularisation
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1313
Participants | 229

30. Secondary Outcome: Clinical Cohort ITT - TVR
Description: Any Target lesion revascularisation
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1277
Participants | 305

31. Secondary Outcome: Clinical Cohort ITT - TVR
Description: Any Target lesion revascularisation
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1242
Participants | 350

32. Secondary Outcome: Clinical Cohort ITT - TVR
Description: Any Target lesion revascularisation
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1386
Participants | 56

33. Secondary Outcome: Clinical Cohort ITT - Time to All-cause Mortality Through 60 Months Post-index Procedure.
Description: All-cause mortality is reported by using the survival estimate of all cause mortality through 60 months
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: percentage of survival
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1406
percentage of survival | 80.5 [78.2 to 82.6]

34. Secondary Outcome: Clinical Cohort ITT - Primary Sustained Clinical Improvement
Description: Primary sustained clinical improvement is defined as sustained upward shift of at least 1 category on Rutherford classification as compared to baseline without the need for repeated TLR or surgical revascularization in amputation-free surviving subjects
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1235
Participants | 1068

35. Secondary Outcome: Clinical Cohort ITT - Primary Sustained Clinical Improvement
Description: as for outcome 34
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1183
Participants | 959

36. Secondary Outcome: Clinical Cohort ITT - Primary Sustained Clinical Improvement
Description: as for outcome 34
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1073
Participants | 745

37. Secondary Outcome: Clinical Cohort ITT - Primary Sustained Clinical Improvement
Description: as for outcome 34
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1009
Participants | 606

38. Secondary Outcome: Clinical Cohort ITT - Secondary Sustained Clinical Improvement
Description: Secondary sustained clinical improvement is defined as sustained upward shift of at least 1 category on Rutherford classification as compared to baseline including the need for repeated TLR or surgical revascularization in amputation-free surviving subjects.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1230
Participants | 1105

39. Secondary Outcome: Clinical Cohort ITT - Secondary Sustained Clinical Improvement
Description: as for outcome 38
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1168
Participants | 1019

40. Secondary Outcome: Clinical Cohort ITT - Secondary Sustained Clinical Improvement
Description: as for outcome 38
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1033
Participants | 876

41. Secondary Outcome: Clinical Cohort ITT - Secondary Sustained Clinical Improvement
Description: as for outcome 38
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 940
Participants | 762

42. Secondary Outcome: Clinical Cohort ITT - Immediate Hemodynamic Improvement at Post-index Procedure
Description: Immediate hemodynamic improvement is defined as an ABI improvement of ≥ 0.1 or to an ABI ≥ 0.9
Time Frame: Post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1225
Participants | 1086

43. Secondary Outcome: Clinical Cohort ITT - Sustained Hemodynamic Improvement
Description: Sustained hemodynamic improvement is defined as persistent improvement of ABI- values with ≥ 0.1 as compared to baseline values or to an ABI ≥ 0.9 throughout follow-up without the need for repeated TLR or surgical revascularization in amputation-free surviving subjects.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1114
Participants | 908

44. Secondary Outcome: Clinical Cohort ITT - Sustained Hemodynamic Improvement
Description: as for outcome 43
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1088
Participants | 797

45. Secondary Outcome: Clinical Cohort ITT - Sustained Hemodynamic Improvement
Description: as for outcome 43
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 986
Participants | 584

46. Secondary Outcome: Clinical Cohort ITT - Sustained Hemodynamic Improvement
Description: as for outcome 43
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 900
Participants | 437

47. Secondary Outcome: Clinical Cohort ITT - Walking Impairment Evaluation by Walking Impairment Questionnaire (WIQ)
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1141
percentage of impairment | 79.7 (29.0)

48. Secondary Outcome: Clinical Cohort ITT - Walking Impairment Evaluation by Walking Impairment Questionnaire (WIQ)
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1109
percentage of impairment | 76.2 (30.7)

49. Secondary Outcome: Clinical Cohort ITT - Walking Impairment Evaluation by Walking Impairment Questionnaire (WIQ)
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 952
percentage of impairment | 75.1 (30.9)

50. Secondary Outcome: Clinical Cohort ITT - Walking Impairment Evaluation by Walking Impairment Questionnaire (WIQ)
Time Frame: 36 Months
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 831
percentage of impairment | 74.4 (30.6)

51. Secondary Outcome: Clinical Cohort ITT - Health Related Quality of Life Scores (EQ5D Index)
Description: The total EQ-5D-3L UK Index Score was computed using the algorithm specified by the EuroQol Research Foundation with possible values ranging from -0.594 to 1 where higher values are better.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1154
score on a scale | 0.8124 (0.2323)

52. Secondary Outcome: Clinical Cohort ITT - Health Related Quality of Life Scores (EQ5D Index)
Description: as for outcome 51
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1114
score on a scale | 0.7970 (0.2413)

53. Secondary Outcome: Clinical Cohort ITT - Health Related Quality of Life Scores (EQ5D Index)
Description: as for outcome 51
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 964
score on a scale | 0.7744 (0.2551)

54. Secondary Outcome: Clinical Cohort ITT - Health Related Quality of Life Scores (EQ5D Index)
Description: as for outcome 51
Time Frame: 36 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 837
score on a scale | 0.7629 (0.2641)

55. Secondary Outcome: Clinical Cohort ITT - Procedural Success
Description: Procedural Success is defined as residual stenosis of ≤ 50% (non-stented subjects) or ≤ 30% (stented subjects) by visual estimate
Time Frame: at procedure
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1406
Number analyzed (lesions) | 1761
lesions | 1750

56. Secondary Outcome: Imaging Cohort ITT - Duplex-defined Binary Restenosis (PSVR > 2.0) of the Target Lesion
Time Frame: at 12 months, or at the time of re-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Imaging Cohort ITT
Number analyzed (Participants) | 252
Participants | 111

57. Secondary Outcome: Imaging Cohort ITT - Duplex-defined Binary Restenosis (PSVR > 3.4) of the Target Lesion
Time Frame: At 12 months, or at the time of re-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Imaging Cohort ITT
Number analyzed (Participants) | 308
Participants | 71

58. Secondary Outcome: 150mm DEB ITT Cohort - MAEs
Description: as for outcome 15
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 114
Participants
  MAEs | 0
  Death | 0
  CD-TVR | 0
  Major Target Limb Amputation | 0
  Thrombosis at Target Lesion Site | 0

59. Secondary Outcome: 150mm DEB ITT Cohort - MAEs
Description: Major Adverse Events (MAE) defined as all-cause death, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants
  MAEs | 6
  Death | 1
  CD-TVR | 5
  Major Target Limb Amputation | 0
  Thrombosis at Target Lesion Site | 1

60. Secondary Outcome: 150mm DEB ITT Cohort - MAEs
Description: Major Adverse Events (MAE) defined as all-cause death, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site at 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants
  MAEs | 9
  Death | 2
  CD-TVR | 7
  Major Target Limb Amputation | 0
  Thrombosis at Target Lesion Site | 1

61. Secondary Outcome: 150mm DEB ITT Cohort - MAEs
Description: Major Adverse Events (MAE) defined as all-cause death, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site at 24 months.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 110
Participants
  MAEs | 22
  Death | 6
  CD-TVR | 17
  Major Target Limb Amputation | 1
  Thrombosis at Target Lesion Site | 2

62. Secondary Outcome: 150mm DEB ITT Cohort - MAEs
Description: Major Adverse Events (MAE) defined as all-cause death, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site at 36 months.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 107
Participants
  MAEs | 37
  Death | 13
  CD-TVR | 26
  Major Target Limb Amputation | 1
  Thrombosis at Target Lesion Site | 2

63. Secondary Outcome: 150mm DEB ITT Cohort - MAEs
Description: Major Adverse Events (MAE) defined as all-cause death, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site at 48 months.
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 106
Participants
  MAEs | 45
  Death | 18
  CD-TVR | 29
  Major Target Limb Amputation | 1
  Thrombosis at Target Lesion Site | 3

64. Secondary Outcome: 150mm DEB ITT Cohort - MAEs
Description: Major Adverse Events (MAE) defined as all-cause death, clinically-driven TVR, major target limb amputation, thrombosis at the target lesion site at 60 months.
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants
  MAEs | 47
  Death | 20
  CD-TVR | 30
  Major Target Limb Amputation | 1
  Thrombosis at Target Lesion Site | 3

65. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 114
Participants | 0

66. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 4

67. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 110
Participants | 16

68. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 107
Participants | 25

69. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 106
Participants | 27

70. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TLR
Description: as for outcome 11
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants | 28

71. Secondary Outcome: 150mm DEB ITT Cohort - TLR
Description: Any Target lesion revascularisation
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 5

72. Secondary Outcome: 150mm DEB ITT Cohort - TLR
Description: Any Target lesion revascularisation
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 7

73. Secondary Outcome: 150mm DEB ITT Cohort - TLR
Description: Any Target lesion revascularisation
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 110
Participants | 17

74. Secondary Outcome: 150mm DEB ITT Cohort - TLR
Description: Any Target lesion revascularisation
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 107
Participants | 26

75. Secondary Outcome: 150mm DEB ITT Cohort - TLR
Description: Any Target lesion revascularisation
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 106
Participants | 28

76. Secondary Outcome: 150mm DEB ITT Cohort - TLR
Description: Any Target lesion revascularisation
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants | 29

77. Secondary Outcome: 150mm DEB ITT Cohort - TVR
Description: Any Target lesion revascularisation
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 6

78. Secondary Outcome: 150mm DEB ITT Cohort - TVR
Description: Any Target lesion revascularisation
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 8

79. Secondary Outcome: 150mm DEB ITT Cohort - TVR
Description: Any Target lesion revascularisation
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 110
Participants | 18

80. Secondary Outcome: 150mm DEB ITT Cohort - TVR
Description: Any Target lesion revascularisation
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 107
Participants | 27

81. Secondary Outcome: 150mm DEB ITT Cohort - TVR
Description: Any Target lesion revascularisation
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 106
Participants | 30

82. Secondary Outcome: 150mm DEB ITT Cohort - TVR
Description: Any Target lesion revascularisation
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants | 31

83. Secondary Outcome: 150mm DEB ITT Cohort - Time to First Clinically-driven TLR (Days)
Time Frame: 60 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 28
Days | 622.2 (352.8)

84. Secondary Outcome: 150mm DEB ITT Cohort - Time to All-cause Mortality Through 60 Months Post-index Procedure.
Description: All-cause mortality is reported by using the survival estimate of all-cause mortality through 60 months
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: percentage of survival
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 116
percentage of survival | 81.1 [72.2 to 87.3]

85. Secondary Outcome: 150mm DEB ITT Cohort - Primary Sustained Clinical Improvement
Description: as for outcome 34
Time Frame: 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 107
Participants | 97

86. Secondary Outcome: 150mm DEB ITT Cohort - Primary Sustained Clinical Improvement
Description: as for outcome 34
Time Frame: 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants | 87

87. Secondary Outcome: 150mm DEB ITT Cohort - Primary Sustained Clinical Improvement
Description: as for outcome 34
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 96
Participants | 68

88. Secondary Outcome: 150mm DEB ITT Cohort - Primary Sustained Clinical Improvement
Description: as for outcome 34
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 92
Participants | 62

89. Secondary Outcome: 150mm DEB ITT Cohort - Secondary Sustained Clinical Improvement
Description: as for outcome 38
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mm DEB ITT Cohort
Number analyzed (Participants) | 106
Participants | 101

90. Secondary Outcome: 150mm DEB ITT Cohort - Secondary Sustained Clinical Improvement
Description: as for outcome 38
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 101
Participants | 90

91. Secondary Outcome: 150mm DEB ITT Cohort - Secondary Sustained Clinical Improvement
Description: as for outcome 38
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 94
Participants | 76

92. Secondary Outcome: 150mm DEB ITT Cohort - Secondary Sustained Clinical Improvement
Description: as for outcome 38
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 89
Participants | 74

93. Secondary Outcome: 150mm DEB ITT Cohort - Immediate Hemodynamic Improvement at Post-index Procedure
Description: Immediate hemodynamic improvement is defined as an ABI improvement of ≥ 0.1 or to an ABI ≥ 0.9
Time Frame: Post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants | 90

94. Secondary Outcome: 150mm DEB ITT Cohort - Sustained Hemodynamic Improvement
Description: as for outcome 43
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 94
Participants | 78

95. Secondary Outcome: 150mm DEB ITT Cohort - Sustained Hemodynamic Improvement
Description: as for outcome 43
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 88
Participants | 72

96. Secondary Outcome: 150mm DEB ITT Cohort - Sustained Hemodynamic Improvement
Description: as for outcome 43
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 85
Participants | 52

97. Secondary Outcome: 150mm DEB ITT Cohort - Sustained Hemodynamic Improvement
Description: as for outcome 43
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 79
Participants | 43

98. Secondary Outcome: 150mm DEB ITT Cohort - Walking Impairment Evaluation by Walking Impairment Questionnaire (WIQ)
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 92
percentage of impairment | 85.9 (23.5)

99. Secondary Outcome: 150mm DEB ITT Cohort - Walking Impairment Evaluation by Walking Impairment Questionnaire (WIQ)
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 86
percentage of impairment | 78.5 (27.4)

100. Secondary Outcome: 150mm DEB ITT Cohort - Walking Impairment Evaluation by Walking Impairment Questionnaire (WIQ)
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 83
percentage of impairment | 77.4 (27.8)

101. Secondary Outcome: 150mm DEB ITT Cohort - Walking Impairment Evaluation by Walking Impairment Questionnaire (WIQ)
Time Frame: 36 Months
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 71
percentage of impairment | 78.5 (25.8)

102. Secondary Outcome: 150mm DEB ITT Cohort - Health Related Quality of Life Scores (EQ5D Index)
Description: as for outcome 51
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 92
score on a scale | 0.8463 (0.1771)

103. Secondary Outcome: 150mm DEB ITT Cohort - Health Related Quality of Life Scores (EQ5D Index)
Description: as for outcome 51
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 86
score on a scale | 0.8257 (0.1853)

104. Secondary Outcome: 150mm DEB ITT Cohort - Health Related Quality of Life Scores (EQ5D Index)
Description: as for outcome 51
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 85
score on a scale | 0.7858 (0.2215)

105. Secondary Outcome: 150mm DEB ITT Cohort - Health Related Quality of Life Scores (EQ5D Index)
Description: as for outcome 51
Time Frame: 36 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 78
score on a scale | 0.8278 (0.2003)

106. Secondary Outcome: 150mm DEB ITT Cohort - Device Success
Description: as for outcome 8
Time Frame: Index-procedure
Measure: Count of Units; unit: Admiral™ Drug-Eluting Balloon
Units Other Than Participants: Admiral™ Drug-Eluting Balloon
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 116
Number analyzed (Admiral™ Drug-Eluting Balloon) | 233
Admiral™ Drug-Eluting Balloon | 231

107. Secondary Outcome: 150mm DEB ITT Cohort - Procedural Success
Description: as for outcome 55
Time Frame: at procedure
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 116
Number analyzed (lesions) | 130
lesions | 130

108. Secondary Outcome: 150mm DEB ITT Cohort - Clinical Success
Description: as for outcome 9
Time Frame: prior to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 116
Participants | 115

109. Secondary Outcome: Clinical Cohort ITT - All-cause Mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1403
Participants | 3

110. Secondary Outcome: Clinical Cohort ITT - All-cause Mortality
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1386
Participants | 23

111. Secondary Outcome: Clinical Cohort ITT - All-cause Mortality
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1361
Participants | 49

112. Secondary Outcome: Clinical Cohort ITT - All-cause Mortality
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1313
Participants | 101

113. Secondary Outcome: Clinical Cohort ITT - All-cause Mortality
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1277
Participants | 147

114. Secondary Outcome: Clinical Cohort ITT - All-cause Mortality
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1242
Participants | 196

115. Secondary Outcome: Clinical Cohort ITT - All-cause Mortality
Description: The difference in death count calculation between the compliance table (participant flow: 253 deaths) and the event table (244 deaths) is explained as follow:
  1. Calendar days (365/year) is used for compliance table whereas 360-day annual cutoff is used for event rate calculation
  2. Compliance table used visit window as specified by protocol (60 days for 5-year follow-up) whereas, not window is used for event rate calculation
  3. Nine patients died between 1801 and 1885 (1825 + 60) and were therefore not included in the 5-year death rate summary but were included in the compliance summary for patients that died through the upper window of the 60 month visit.
  4. The denominator of 1215 for 1800-day event rate includes those who had an event within 1800 days and those who did not have any event but had at least 1740 days of follow-up (1740 is the low bound of the 60-day visit window from the target day of 1800)
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1215
Participants | 244

116. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TVR
Description: Clinically-driven TVR is defined as any re-intervention within the target vessel due to symptoms or drop of ABI of ≥ 20% or > 0.15 when compared to post-index procedure baseline ABI.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1403
Participants | 13

117. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1386
Participants | 54

118. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1361
Participants | 107

119. Secondary Outcome: Clinical Clinical Cohort ITT - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1313
Participants | 224

120. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1277
Participants | 298

121. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1242
Participants | 342

122. Secondary Outcome: Clinical Cohort ITT - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1215
Participants | 381

123. Secondary Outcome: Clinical Cohort ITT - Major Target Limb Amputation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1403
Participants | 0

124. Secondary Outcome: Clinical Cohort ITT - Major Target Limb Amputation
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1386
Participants | 3

125. Secondary Outcome: Clinical Cohort ITT - Major Target Limb Amputation
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1361
Participants | 3

126. Secondary Outcome: Clinical Cohort ITT - Major Target Limb Amputation
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1313
Participants | 57

127. Secondary Outcome: Clinical Cohort ITT - Major Target Limb Amputation
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1277
Participants | 12

128. Secondary Outcome: Clinical Cohort ITT - Major Target Limb Amputation
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1242
Participants | 15

129. Secondary Outcome: Clinical Cohort ITT - Major Target Limb Amputation
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Cohort ITT
Number analyzed (Participants) | 1215
Participants | 19

130. Secondary Outcome: 150mm DEB ITT Cohort - All-cause Mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 114
Participants | 0

131. Secondary Outcome: 150mm DEB ITT Cohort - All-cause Mortality
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 1

132. Secondary Outcome: 150mm DEB ITT Cohort - All-cause Mortality
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 2

133. Secondary Outcome: 150mm DEB ITT Cohort - All-cause Mortality
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 110
Participants | 6

134. Secondary Outcome: 150mm DEB ITT Cohort - All-cause Mortality
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 107
Participants | 13

135. Secondary Outcome: 150mm DEB ITT Cohort - All-cause Mortality
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 106
Participants | 18

136. Secondary Outcome: 150mm DEB ITT Cohort - All-cause Mortality
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants | 20

137. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 114
Participants | 0

138. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 5

139. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 7

140. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 110
Participants | 17

141. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 107
Participants | 26

142. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 106
Participants | 29

143. Secondary Outcome: 150mm DEB ITT Cohort - Clinically-driven TVR
Description: as for outcome 116
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants | 30

144. Secondary Outcome: 150mm DEB ITT Cohort - Major Target Limb Amputation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 114
Participants | 0

145. Secondary Outcome: 150mm DEB ITT Cohort - Major Target Limb Amputation
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 0

146. Secondary Outcome: 150mm DEB ITT Cohort - Major Target Limb Amputation
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 112
Participants | 0

147. Secondary Outcome: 150mm DEB ITT Cohort - Major Target Limb Amputation
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 110
Participants | 1

148. Secondary Outcome: 150mm DEB ITT Cohort - Major Target Limb Amputation
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 107
Participants | 1

149. Secondary Outcome: 150mm DEB ITT Cohort - Major Target Limb Amputation
Time Frame: 48 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 106
Participants | 1

150. Secondary Outcome: 150mm DEB ITT Cohort - Major Target Limb Amputation
Time Frame: 60 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 102
Participants | 1

151. Secondary Outcome: 150mm DEB ITT Cohort - Time to First Clinically-driven TLR (Days)
Time Frame: 60 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 150mm DEB ITT Cohort
Number analyzed (Participants) | 28
Days | 622.2 (352.8)

ADVERSE EVENTS:
Time Frame: 60 Months
Groups:
- Clinical Cohort 60M: Events through the entire 60 months follow-up period are included
Arm/Group | Clinical Cohort 60M
All-Cause Mortality (participants affected / at risk) | 253/1406
Serious Adverse Events (participants affected / at risk) | 1074/1406
Other Adverse Events (participants affected / at risk) | 287/1406
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Cohort 60M (N=1406)
Anaemia (Blood and lymphatic system disorders) | 23 (24)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 5 (5)
Haemorrhagic Disorder (Blood and lymphatic system disorders) | 2 (2)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 1 (1)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Acute Coronary Syndrome (Cardiac disorders) | 6 (6)
Acute Myocardial Infarction (Cardiac disorders) | 52 (57)
Angina Pectoris (Cardiac disorders) | 34 (37)
Angina Unstable (Cardiac disorders) | 20 (22)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 8 (9)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 4 (4)
Atrial Fibrillation (Cardiac disorders) | 31 (34)
Atrial Flutter (Cardiac disorders) | 6 (6)
Atrial Thrombosis (Cardiac disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 5 (5)
Atrioventricular Block Complete (Cardiac disorders) | 3 (3)
Atrioventricular Block Second Degree (Cardiac disorders) | 1 (1)
Atrioventricular Dissociation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 8 (8)
Bundle Branch Block Left (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 19 (19)
Cardiac Disorder (Cardiac disorders) | 2 (2)
Cardiac Failure (Cardiac disorders) | 53 (66)
Cardiac Failure Acute (Cardiac disorders) | 6 (6)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 3 (3)
Cardiac Valve Disease (Cardiac disorders) | 2 (2)
Cardio-Respiratory Arrest (Cardiac disorders) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 5 (5)
Cardiomegaly (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (2)
Cardiopulmonary Failure (Cardiac disorders) | 4 (4)
Cardiovascular Insufficiency (Cardiac disorders) | 1 (1)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 51 (54)
Coronary Artery Insufficiency (Cardiac disorders) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 6 (7)
Coronary Artery Stenosis (Cardiac disorders) | 26 (32)
Coronary Artery Thrombosis (Cardiac disorders) | 1 (1)
Diastolic Dysfunction (Cardiac disorders) | 1 (1)
Heart Valve Incompetence (Cardiac disorders) | 2 (2)
Hypertensive Cardiomyopathy (Cardiac disorders) | 1 (1)
Hypertensive Heart Disease (Cardiac disorders) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 3 (3)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Left Ventricular Failure (Cardiac disorders) | 1 (1)
Low Cardiac Output Syndrome (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 4 (4)
Mitral Valve Stenosis (Cardiac disorders) | 1 (1)
Myocardial Fibrosis (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 25 (25)
Myocardial Ischaemia (Cardiac disorders) | 8 (8)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Rhythm Idioventricular (Cardiac disorders) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 3 (3)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Stress Cardiomyopathy (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 3 (3)
Trifascicular Block (Cardiac disorders) | 1 (1)
Ventricle Rupture (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Congenital Arterial Malformation (Congenital, familial and genetic disorders) | 1 (1)
Gastrointestinal Angiodysplasia (Congenital, familial and genetic disorders) | 2 (2)
Phimosis (Congenital, familial and genetic disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 9 (10)
Vertigo Positional (Ear and labyrinth disorders) | 2 (2)
Goitre (Endocrine disorders) | 2 (2)
Hyperparathyroidism Tertiary (Endocrine disorders) | 1 (1)
Amaurosis Fugax (Eye disorders) | 1 (1)
Blindness Unilateral (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 18 (25)
Cataract Cortical (Eye disorders) | 1 (1)
Dacryostenosis Acquired (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Lens Dislocation (Eye disorders) | 1 (1)
Macular Degeneration (Eye disorders) | 2 (2)
Retinal Artery Occlusion (Eye disorders) | 1 (1)
Retinal Detachment (Eye disorders) | 2 (2)
Visual Impairment (Eye disorders) | 2 (3)
Vitreous Adhesions (Eye disorders) | 1 (1)
Vitreous Haemorrhage (Eye disorders) | 2 (3)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (4)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (5)
Abdominal Symptom (Gastrointestinal disorders) | 1 (1)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 1 (1)
Acute Abdomen (Gastrointestinal disorders) | 2 (2)
Anal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Anal Skin Tags (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 5 (5)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1)
Colonic Polyp (Gastrointestinal disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 3 (3)
Dental Caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Enteritis (Gastrointestinal disorders) | 2 (2)
Erosive Duodenitis (Gastrointestinal disorders) | 1 (1)
Faecal Vomiting (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 2 (2)
Food Poisoning (Gastrointestinal disorders) | 1 (1)
Gastric Haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastric Perforation (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 4 (4)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 3 (3)
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 7 (8)
Gastritis Erosive (Gastrointestinal disorders) | 2 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 15 (15)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 4 (4)
Inguinal Hernia (Gastrointestinal disorders) | 9 (9)
Intestinal Ischaemia (Gastrointestinal disorders) | 5 (5)
Intestinal Obstruction (Gastrointestinal disorders) | 2 (2)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Intestinal Polyp (Gastrointestinal disorders) | 1 (1)
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 1 (1)
Jejunal Ulcer (Gastrointestinal disorders) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 2 (2)
Lumbar Hernia (Gastrointestinal disorders) | 1 (1)
Malignant Dysphagia (Gastrointestinal disorders) | 1 (1)
Mechanical Ileus (Gastrointestinal disorders) | 1 (1)
Mesenteric Artery Stenosis (Gastrointestinal disorders) | 6 (7)
Oesophageal Achalasia (Gastrointestinal disorders) | 1 (1)
Oesophageal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 3 (4)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 2 (2)
Pancreatitis Chronic (Gastrointestinal disorders) | 2 (2)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 4 (4)
Rectal Polyp (Gastrointestinal disorders) | 1 (1)
Reflux Oesophagitis (Gastrointestinal disorders) | 3 (3)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 2 (2)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 3 (3)
Sigmoiditis (Gastrointestinal disorders) | 1 (1)
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Spigelian Hernia (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 2 (2)
Umbilical Hernia (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Cardiac Death (General disorders) | 3 (3)
Chest Discomfort (General disorders) | 2 (2)
Chest Pain (General disorders) | 12 (14)
Death (General disorders) | 55 (55)
Device Breakage (General disorders) | 3 (3)
Device Dislocation (General disorders) | 2 (2)
Device Malfunction (General disorders) | 1 (1)
Device Occlusion (General disorders) | 45 (49)
Euthanasia (General disorders) | 1 (1)
Exercise Tolerance Decreased (General disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)
General Physical Health Deterioration (General disorders) | 4 (4)
Hernia (General disorders) | 1 (1)
Hernia Obstructive (General disorders) | 2 (2)
Hyperplasia (General disorders) | 2 (2)
Impaired Healing (General disorders) | 9 (13)
Inflammation (General disorders) | 1 (1)
Infusion Site Extravasation (General disorders) | 1 (1)
Malaise (General disorders) | 4 (4)
Multi-Organ Failure (General disorders) | 5 (5)
Oedema Peripheral (General disorders) | 3 (3)
Puncture Site Haemorrhage (General disorders) | 1 (1)
Sudden Cardiac Death (General disorders) | 1 (1)
Sudden Death (General disorders) | 1 (1)
Thrombosis In Device (General disorders) | 9 (12)
Vessel Puncture Site Discharge (General disorders) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 3 (3)
Vessel Puncture Site Haemorrhage (General disorders) | 7 (7)
Vessel Puncture Site Reaction (General disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 3 (3)
Cholangitis Acute (Hepatobiliary disorders) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 4 (4)
Cholecystitis Acute (Hepatobiliary disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 6 (6)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Gallbladder Necrosis (Hepatobiliary disorders) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Liver Disorder (Hepatobiliary disorders) | 2 (2)
Anaphylactic Reaction (Immune system disorders) | 2 (3)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Abscess (Infections and infestations) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Appendicitis Perforated (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bone Abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Bronchopneumonia (Infections and infestations) | 4 (4)
Cellulitis (Infections and infestations) | 9 (10)
Clostridium Difficile Colitis (Infections and infestations) | 2 (3)
Cystitis (Infections and infestations) | 1 (1)
Device Related Infection (Infections and infestations) | 5 (6)
Diabetic Gangrene (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3)
Endocarditis (Infections and infestations) | 2 (2)
Enterococcal Infection (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 13 (13)
Febrile Infection (Infections and infestations) | 1 (1)
Fungal Infection (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 19 (21)
Gastroenteritis (Infections and infestations) | 3 (4)
Gastroenteritis Viral (Infections and infestations) | 1 (1)
Gastrointestinal Candidiasis (Infections and infestations) | 1 (1)
Graft Infection (Infections and infestations) | 2 (2)
Groin Abscess (Infections and infestations) | 2 (2)
Groin Infection (Infections and infestations) | 2 (2)
Haematoma Infection (Infections and infestations) | 2 (2)
Helicobacter Gastritis (Infections and infestations) | 1 (1)
Hepatic Infection (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 3 (3)
Herpes Zoster Infection Neurological (Infections and infestations) | 1 (1)
Herpes Zoster Ophthalmic (Infections and infestations) | 1 (1)
Infected Lymphocele (Infections and infestations) | 1 (1)
Infected Skin Ulcer (Infections and infestations) | 4 (4)
Infection (Infections and infestations) | 8 (8)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 4 (4)
Kidney Infection (Infections and infestations) | 1 (1)
Localised Infection (Infections and infestations) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2)
Lung Infection (Infections and infestations) | 2 (2)
Necrotising Fasciitis (Infections and infestations) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 11 (12)
Osteomyelitis Chronic (Infections and infestations) | 1 (1)
Periorbital Cellulitis (Infections and infestations) | 1 (1)
Peritoneal Abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 70 (85)
Post Procedural Infection (Infections and infestations) | 1 (1)
Postoperative Abscess (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 6 (7)
Prostatic Abscess (Infections and infestations) | 1 (1)
Pseudomembranous Colitis (Infections and infestations) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 7 (7)
Pyelonephritis (Infections and infestations) | 2 (2)
Pyothorax (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 10 (10)
Septic Shock (Infections and infestations) | 4 (4)
Severe Acute Respiratory Syndrome (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 12 (13)
Urosepsis (Infections and infestations) | 6 (7)
Viral Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 8 (8)
Wound Infection Bacterial (Infections and infestations) | 1 (1)
Wound Infection Staphylococcal (Infections and infestations) | 2 (3)
Wound Sepsis (Infections and infestations) | 2 (3)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 (1)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 5 (5)
Anastomotic Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Arterial Injury (Injury, poisoning and procedural complications) | 2 (2)
Arterial Restenosis (Injury, poisoning and procedural complications) | 143 (204)
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Chemical Peritonitis (Injury, poisoning and procedural complications) | 1 (1)
Colon Injury (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 4 (5)
Drug Toxicity (Injury, poisoning and procedural complications) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 6 (6)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 3 (3)
Femoral Nerve Injury (Injury, poisoning and procedural complications) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 6 (6)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 3 (3)
Foreign Body (Injury, poisoning and procedural complications) | 1 (1)
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 2 (2)
Hip Fracture (Injury, poisoning and procedural complications) | 3 (3)
Humerus Fracture (Injury, poisoning and procedural complications) | 3 (4)
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 87 (113)
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 3 (3)
Incisional Hernia (Injury, poisoning and procedural complications) | 2 (3)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 4 (4)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1)
Multiple Injuries (Injury, poisoning and procedural complications) | 1 (1)
Nerve Injury (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1)
Peripheral Arterial Reocclusion (Injury, poisoning and procedural complications) | 40 (52)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 1 (1)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 1 (3)
Post Procedural Complication (Injury, poisoning and procedural complications) | 3 (3)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Post Procedural Swelling (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Pubis Fracture (Injury, poisoning and procedural complications) | 1 (1)
Radiation Oesophagitis (Injury, poisoning and procedural complications) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 3 (3)
Rib Fracture (Injury, poisoning and procedural complications) | 3 (4)
Shunt Occlusion (Injury, poisoning and procedural complications) | 1 (1)
Shunt Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 2 (2)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 (2)
Spinal Fracture (Injury, poisoning and procedural complications) | 2 (2)
Sternal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 5 (5)
Tendon Rupture (Injury, poisoning and procedural complications) | 2 (2)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 3 (3)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Ulna Fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2 (2)
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 1 (1)
Vascular Graft Complication (Injury, poisoning and procedural complications) | 11 (11)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 20 (23)
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 9 (13)
Vascular Procedure Complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 33 (36)
Venous Injury (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 6 (6)
Wound Complication (Injury, poisoning and procedural complications) | 2 (2)
Wound Decomposition (Injury, poisoning and procedural complications) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Wound Necrosis (Injury, poisoning and procedural complications) | 2 (2)
Arteriogram Coronary (Investigations) | 1 (1)
Blood Creatinine Increased (Investigations) | 5 (5)
Blood Glucose Abnormal (Investigations) | 1 (1)
Blood Glucose Fluctuation (Investigations) | 1 (1)
Blood Glucose Increased (Investigations) | 1 (1)
Blood Sodium Decreased (Investigations) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1)
Chest X-Ray Abnormal (Investigations) | 1 (1)
Clostridium Test Positive (Investigations) | 1 (1)
Haemoglobin Decreased (Investigations) | 4 (4)
International Normalised Ratio Increased (Investigations) | 2 (2)
Investigation (Investigations) | 2 (2)
Scan Abnormal (Investigations) | 1 (1)
Transplant Evaluation (Investigations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 7 (7)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 4 (4)
Diabetic Foot (Metabolism and nutrition disorders) | 10 (11)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6)
Insulin Resistance (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1)
Metabolic Syndrome (Metabolism and nutrition disorders) | 1 (1)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 13 (13)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 (2)
Fistula (Musculoskeletal and connective tissue disorders) | 2 (2)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 3 (3)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 10 (10)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 10 (10)
Meniscal Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nodule On Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 23 (24)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 11 (11)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 3 (3)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 6 (7)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2)
Systemic Sclerosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 3 (3)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 2 (5)
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign Spleen Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bladder Transitional Cell Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bone Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Carcinoid Tumour Of The Caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carcinoma In Situ Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Laryngeal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lentigo Maligna Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Lung Adenocarcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Adenocarcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant Neoplasm Of Uterine Adnexa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Metastases To Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mixed Hepatocellular Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neoplasm Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's Lymphoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Oral Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Penis Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Respiratory Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Salivary Gland Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Undifferentiated Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered State Of Consciousness (Nervous system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Basal Ganglia Haemorrhage (Nervous system disorders) | 1 (1)
Basal Ganglia Infarction (Nervous system disorders) | 1 (1)
Brain Oedema (Nervous system disorders) | 1 (1)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 33 (38)
Carpal Tunnel Syndrome (Nervous system disorders) | 8 (11)
Cerebral Artery Occlusion (Nervous system disorders) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 5 (5)
Cerebral Infarction (Nervous system disorders) | 4 (4)
Cerebral Ischaemia (Nervous system disorders) | 1 (1)
Cerebral Thrombosis (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 29 (30)
Cervical Root Pain (Nervous system disorders) | 1 (1)
Coordination Abnormal (Nervous system disorders) | 1 (1)
Critical Illness Polyneuropathy (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 3 (3)
Dementia Alzheimer's Type (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Embolic Cerebral Infarction (Nervous system disorders) | 2 (2)
Embolic Stroke (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 3 (4)
Facial Palsy (Nervous system disorders) | 2 (2)
Guillain-Barre Syndrome (Nervous system disorders) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 3 (3)
Intracranial Aneurysm (Nervous system disorders) | 1 (1)
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 12 (12)
Lacunar Infarction (Nervous system disorders) | 1 (1)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (2)
Neuropathy Peripheral (Nervous system disorders) | 1 (1)
Normal Pressure Hydrocephalus (Nervous system disorders) | 1 (1)
Parkinson's Disease (Nervous system disorders) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1)
Post-Traumatic Headache (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Reversible Ischaemic Neurological Deficit (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 3 (3)
Speech Disorder (Nervous system disorders) | 1 (1)
Spinal Claudication (Nervous system disorders) | 1 (1)
Status Epilepticus (Nervous system disorders) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 14 (14)
Thoracic Outlet Syndrome (Nervous system disorders) | 1 (1)
Thrombotic Stroke (Nervous system disorders) | 1 (1)
Toxic Neuropathy (Nervous system disorders) | 1 (1)
Transient Global Amnesia (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 10 (10)
Vascular Encephalopathy (Nervous system disorders) | 1 (1)
Alcohol Abuse (Psychiatric disorders) | 1 (3)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Behavioural And Psychiatric Symptoms Of Dementia (Psychiatric disorders) | 1 (1)
Breathing-Related Sleep Disorder (Psychiatric disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 7 (7)
Depression (Psychiatric disorders) | 4 (5)
Disorientation (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Mood Disorder Due To A General Medical Condition (Psychiatric disorders) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 2 (2)
Azotaemia (Renal and urinary disorders) | 1 (1)
Bladder Prolapse (Renal and urinary disorders) | 1 (1)
Bladder Tamponade (Renal and urinary disorders) | 1 (1)
Cystitis Haemorrhagic (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Nephropathy Toxic (Renal and urinary disorders) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 3 (3)
Renal Colic (Renal and urinary disorders) | 1 (1)
Renal Cyst (Renal and urinary disorders) | 2 (2)
Renal Disorder (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 17 (17)
Renal Failure Acute (Renal and urinary disorders) | 22 (26)
Renal Failure Chronic (Renal and urinary disorders) | 8 (8)
Renal Impairment (Renal and urinary disorders) | 4 (4)
Stress Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Ureteric Stenosis (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 5 (5)
Urinary Tract Disorder (Renal and urinary disorders) | 1 (1)
Adnexa Uteri Mass (Reproductive system and breast disorders) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 8 (8)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1)
Endometrial Hypertrophy (Reproductive system and breast disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Pelvic Haematoma (Reproductive system and breast disorders) | 1 (1)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 2 (2)
Prostatic Obstruction (Reproductive system and breast disorders) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 1 (1)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1)
Uterine Prolapse (Reproductive system and breast disorders) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 17 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epiglottic Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal Leukoplakia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung Cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 (3)
Dry Gangrene (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 27 (31)
Abdominal Hernia Repair (Surgical and medical procedures) | 1 (1)
Aortic Aneurysm Repair (Surgical and medical procedures) | 1 (1)
Arterial Stent Insertion (Surgical and medical procedures) | 1 (1)
Arteriovenous Fistula Operation (Surgical and medical procedures) | 2 (2)
Cardiac Pacemaker Battery Replacement (Surgical and medical procedures) | 2 (2)
Cataract Operation (Surgical and medical procedures) | 1 (1)
Central Venous Catheterisation (Surgical and medical procedures) | 1 (1)
Coronary Artery Bypass (Surgical and medical procedures) | 1 (1)
Debridement (Surgical and medical procedures) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Ileostomy Closure (Surgical and medical procedures) | 1 (1)
Implantable Defibrillator Replacement (Surgical and medical procedures) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 2 (3)
Leg Amputation (Surgical and medical procedures) | 2 (2)
Medical Device Change (Surgical and medical procedures) | 1 (1)
Medical Device Removal (Surgical and medical procedures) | 1 (1)
Peripheral Artery Angioplasty (Surgical and medical procedures) | 3 (3)
Peripheral Revascularisation (Surgical and medical procedures) | 3 (4)
Portal Shunt (Surgical and medical procedures) | 1 (2)
Renal Transplant (Surgical and medical procedures) | 1 (1)
Toe Amputation (Surgical and medical procedures) | 1 (1)
Tympanoplasty (Surgical and medical procedures) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (2)
Aortic Aneurysm (Vascular disorders) | 4 (4)
Aortic Aneurysm Rupture (Vascular disorders) | 1 (1)
Aortic Arteriosclerosis (Vascular disorders) | 1 (1)
Aortic Disorder (Vascular disorders) | 1 (1)
Aortic Stenosis (Vascular disorders) | 2 (2)
Arterial Disorder (Vascular disorders) | 1 (1)
Arterial Haemorrhage (Vascular disorders) | 6 (7)
Arterial Rupture (Vascular disorders) | 4 (4)
Arterial Spasm (Vascular disorders) | 1 (1)
Arterial Stenosis (Vascular disorders) | 5 (5)
Arterial Stenosis Limb (Vascular disorders) | 89 (115)
Arterial Thrombosis (Vascular disorders) | 4 (5)
Arterial Thrombosis Limb (Vascular disorders) | 62 (76)
Arteriosclerosis (Vascular disorders) | 4 (4)
Arteriosclerosis Obliterans (Vascular disorders) | 3 (4)
Artery Dissection (Vascular disorders) | 1 (1)
Circulatory Collapse (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Embolism Venous (Vascular disorders) | 1 (1)
Extremity Necrosis (Vascular disorders) | 13 (13)
Femoral Arterial Stenosis (Vascular disorders) | 260 (397)
Femoral Artery Aneurysm (Vascular disorders) | 3 (5)
Femoral Artery Dissection (Vascular disorders) | 4 (4)
Femoral Artery Embolism (Vascular disorders) | 2 (2)
Femoral Artery Occlusion (Vascular disorders) | 137 (170)
Haematoma (Vascular disorders) | 19 (21)
Haemorrhage (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 9 (11)
Hypertensive Crisis (Vascular disorders) | 9 (10)
Hypovolaemic Shock (Vascular disorders) | 2 (2)
Iliac Artery Embolism (Vascular disorders) | 1 (1)
Iliac Artery Occlusion (Vascular disorders) | 10 (11)
Iliac Artery Stenosis (Vascular disorders) | 95 (123)
Iliac Artery Thrombosis (Vascular disorders) | 3 (3)
Intermittent Claudication (Vascular disorders) | 55 (64)
Ischaemia (Vascular disorders) | 1 (1)
Ischaemic Limb Pain (Vascular disorders) | 4 (4)
Leriche Syndrome (Vascular disorders) | 1 (1)
Lymphatic Fistula (Vascular disorders) | 1 (1)
Lymphocele (Vascular disorders) | 2 (2)
Necrosis Ischaemic (Vascular disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 122 (161)
Peripheral Artery Aneurysm (Vascular disorders) | 3 (3)
Peripheral Artery Dissection (Vascular disorders) | 5 (5)
Peripheral Embolism (Vascular disorders) | 13 (13)
Peripheral Ischaemia (Vascular disorders) | 33 (41)
Shock (Vascular disorders) | 1 (1)
Steal Syndrome (Vascular disorders) | 1 (1)
Subclavian Artery Occlusion (Vascular disorders) | 1 (2)
Subclavian Artery Stenosis (Vascular disorders) | 2 (2)
Subclavian Steal Syndrome (Vascular disorders) | 1 (1)
Thromboangiitis Obliterans (Vascular disorders) | 2 (3)
Varicophlebitis (Vascular disorders) | 1 (1)
Varicose Vein (Vascular disorders) | 3 (3)
Vascular Calcification (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Venous Haemorrhage (Vascular disorders) | 1 (1)
Venous Stenosis (Vascular disorders) | 2 (2)
Venous Thrombosis Limb (Vascular disorders) | 2 (2)
Vessel Perforation (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Cohort 60M (N=1406)
Femoral Arterial Stenosis (Vascular disorders) | 142 (175)
Intermittent Claudication (Vascular disorders) | 73 (80)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 72 (85)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less